CLINICAL TRIAL: NCT07309250
Title: Gastrointestinal Transit Time at the Population Level: A Cross-sectional Study
Brief Title: A Study on Gastrointestinal Transit Time at the Population Level
Acronym: GITTPop
Status: Not yet recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Christophe Matthys, Professor, KU Leuven
Other Study IDs: S70908
Record Dates: First submitted 2025-11-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Transit Time
Keywords: Gastrointestinal motility; Baseline study; Reference value
MeSH Terms: interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult participants: Healthy adult participants without serious gastrointestinal diseases
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Participants will consume a regular muffin containing blue dye

SUMMARY:
The goal of this study is to investigate the baseline of gastrointestinal transit time (GITT) and explore its relationship with other health indicators in 932 healthy adult volunteers.

The main questions it aims to answer are:

What are the population-level baseline values for GITT using the blue dye method? How is GITT associated with key physiological parameters including blood metabolic markers, life style, and stool characteristics?

Participants will:

Consume a standardized blue dye muffin after overnight fasting at the research center; Offer a finger prock blood samples for metabolic profiling; Collect stool samples for moisture measurement; Complete detailed questionnaires on diet, lifestyle, and bowel habits; Record the time of first blue stool appearance to determine GITT.

DETAILED DESCRIPTION:
This explorative study is designed as a cross-sectional investigation aimed at establishing population-level reference values for gastrointestinal transit time (GITT). Adult participants from the general population will undergo GITT measurement using the blue-dye method. This muffin contains blue colorant that cannot be absorbed; after ingestion, it passes through the entire gastrointestinal tract and is eventually excreted in feces. Following a two-day lifestyle standardization period (including dietary and activity guidance) to minimize potential confounding effects on gastrointestinal motility, participants will attend a clinical visit where they will ingest a blue muffin. GITT will be determined by measuring both the time interval between ingestion of the blue muffin and the first appearance of blue-colored stool, and the duration from its first appearance to its complete disappearance.

The blue muffin method has been well-established in previous research for GITT assessment. Building upon the methodology developed by Berry et al., we will introduce stricter pre-test condition controls (includes dietary advice and lifestyle recommendations) and optimized the blue muffin formulation.These improvements allow for reliable measurement with a single muffin administration, which has been evaluated through KU Leuven Health Pass in a large sample size(S-70168).

To investigate potential determinants and correlates of GITT, we will collect biochemical parameters, fecal moisture, and resting metabolic rate. Additionally, participants will complete 24-h diet record and health questionnaires assessing bowel movement, physical activity habits, stress levels, sleep quality and hydration condition for subsequent correlation analyses.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old
2. 18.5 kg/m² ≤ BMI ≤ 25 kg/m² or BMI ≥ 30 kg/m² (people with normal weight or obesity)
3. Provision of informed consent to participate.

Exclusion Criteria:

1. Gastrointestinal conditions which may affect nutrient absorption or gastric emptying, including coeliac disease, Crohn's disease, previous resection of the small intestine other than bariatric surgery, gastroparesis;
2. Using medications which effect gastric motility (e.g., domperidone, erythromycin, metoclopramide, prucalopride, opiates, loperamide, …)
3. The ingredients of blue muffins include gluten, nuts, baking powder, sugar, vanilla extract and sunflower oil. Participants with allergies to these ingredients;
4. Current diagnosis of cancer;
5. Advanced organ failure, including chronic kidney disease Stage 5, liver cirrhosis Child-Pugh B or C, intestinal failure, heart failure stage D, or chronic obstructive pulmonary disease stage 4;
6. Immobility;
7. Neuromuscular degenerative conditions associated with muscular atrophy, such as myasthenia gravis, muscular dystrophies, fibromyalgia, or multiple Sclerosis;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers from the Flanders region who volunteered to participate in the research
Sampling Method: Non-Probability Sample
Enrollment: 932 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal transit time | From enrollment to the end of study at 2 weeks
  Calculate the transit time by the recorded muffin consuming time, first blue stool appearance time and last blue stool appearance time

SECONDARY OUTCOMES:
Height (cm) | baseline
  Measured using a height meter, in centimeters.
Weight (kg) | baseline
  Measuring using a scale, in kg.
BMI | baseline
  weight and height will be combined to report BMI in kg/m^2
Blood glucose (mmol/L) | baseline
  Measure blood glucose by CardioChek Plus in mmol/L
Fat mass (kg) | baseline
  Using Bodystat quadscan 4000 to measure fat mass (kg)
Lean body mass(kg) | baseline
  Using Bodystat quadscan 4000 to measure lean body mass (kg)
Fat percentage (%) | baseline
  Using Bodystat quadscan 4000 to measure fat%
Total cholesterol (mmol/L) | baseline
  Measuring by Mission cholesterol Meter in mmol/L
HDL-C (mmol/L) | baseline
  Measuring by Mission cholesterol Meter in mmol/L
LDL-C (mmol/L) | baseline
  Measuring by Mission cholesterol Meter in mmol/L
Triglyceride (mmol/L) | baseline
  Measuring by Mission Cholesterol Meter in mmol/L
Food record | 2 days after study
  Participants record their 24-h diets through smartphone application
Stool form | baseline
  Stool form will be evaluated by Bristol Stool Form Scale, the score is from 1 to 7, with values closer to the middle indicating more ideal stool shape.
Hydration status | baseline
  Hydration status will be rated from 1 to 8 by Urine color chart, with higher numbers indicating that the body needs more water.
Perceived level of stress | baseline
  The10-item Perceived Stress will be used to measures an individual's perceived level of stress over the past month. The total score ranges from 0 to 40. A higher score indicates a greater perceived level of stress.
Sleep quality | baseline
  Pittsburgh Sleep Quality Index will be used to assess subjective sleep quality over the past month. The total score ranges from 0 to 21. A higher score indicates poorer sleep quality.
Activity level | baseline
  The Baecke Physical Activity Questionnaire will be used to assess daily habitual physical activity, with a particular focus on work-related and exercise-related activities. It does not produce a single total score, but rather scores on three dimensions, each typically ranging from 1 to 5. On each dimension, a higher score indicates a higher level of physical activity in that area. Therefore, for assessing activity levels, a higher score is generally better.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Chronic Diseases and Metabolism, Leuven, Flemish Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT07309250/Prot_SAP_000.pdf